CLINICAL TRIAL: NCT03110263
Title: i-Sleep: Internet-based Treatment for Insomnia. A Randomized Controlled Trial
Brief Title: i-Sleep: Internet-based Treatment for Insomnia
Acronym: i-Sleep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: practicality reasons; recruitment slower than expected
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-00295
Record Dates: First submitted 2017-03-28; First posted 2017-04-12 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multicomponent internet-based self-help (Experimental): Multicomponent internet-based self-help
  Interventions: Other: Multicomponent internet-based self-help
- Internet-based sleep restriction (Experimental): Internet-based sleep restriction
  Interventions: Other: Internet-based sleep restriction
- Waiting control group (No Intervention): Access to internet-based intervention after 8-weeks

INTERVENTIONS:
Other: Multicomponent internet-based self-help — Internet-based self-help on the basis of (Perlis, M. L., Jungquist, C., Smith, M. T., & Posner, D., 2006). The self-help program consists of eight text-based sessions and tasks. All participants in the active conditions receive guidance during 8-weeks treatment.
  Arms: Multicomponent internet-based self-help
Other: Internet-based sleep restriction — Internet-based self-help on the basis of (Perlis, M. L., Jungquist, C., Smith, M. T., & Posner, D., 2006). The self-help program consists of five text-based sessions and tasks. All participants in the active conditions receive guidance during 8-weeks treatment.
  Arms: Internet-based sleep restriction

SUMMARY:
In this study, people who suffer from insomnia will be randomized to one of three study conditions. The first group receives a multicomponent internet-based cognitive behavioral self-help intervention. The second group has access to an internet-based self-help sleep restriction intervention. The third group is a waiting control group. In both active conditions additional care or treatment is allowed. The aim of the study is to investigate the effectiveness of a multicomponent internet-based cognitive behavioral self-help intervention as well as a stand-alone internet-based self-help sleep restriction intervention for insomnia symptoms compared to a waiting list. Assessments take place at baseline, and 8-weeks and 6-months post-randomization. After 8 weeks, participants in the waiting control group get access to the internet-based cognitive behavioural self-help intervention and also fill out questionnaires at 6-months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Meet ICSD-3 diagnostic criteria for Insomnia as confirmed by the telephone administered Interview
* Acess to the Internet
* Written informed consent

Exclusion Criteria:

* Physiological Insomnia
* Serious psychiatric co-morbidity that requires alternative treatment including major depression disorder, anxiety disorder, substance dependence, bipolar affective disorder, psychotic illness
* Epilepsy (seizure disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2018-01-07 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline
Insomnia Severity Index (ISI) | 8-weeks
Insomnia Severity Index (ISI) | 6-months

SECONDARY OUTCOMES:
Diagnosis of Insomnia | Baseline, 8-weeks, 6-months
  International Classification of Insomnia Disorders (ICSD-3)
Sleep-diary: Sleep efficiency (SE) | 8-weeks
Sleep-Diary-data | 8-weeks
Dysfunctional Beliefs and Attitudes about Sleep 16 (DBAS-16) | Baseline, 8-weeks, 6-months
Patient satisfaction (ZUF-8) | 8-weeks
Empowerment Scale (ES) | Baseline, 8-weeks, 6-months
EuroQol | Baseline, 8-weeks, 6-months
Usability: Satisfaction with the online program (SUS) | 8-weeks
Pittsburgh Sleep Quality Index (PSQI) | Baseline, 8-weeks, 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berger, PhD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No